CLINICAL TRIAL: NCT00651846
Title: Single Center, Double Blind, Randomized, Crossover Study to Investigate the Impact of the Oral Contraceptive Yasmin (30 µg EE / 3 mg DRSP) Compared to Microgynon (30 µg / 150 LNG) on Hemostasis Parameters in 40 Female Volunteers
Brief Title: Investigate Impact of Yasmin vs Microgynon on Hemostasis Parameters in Healthy Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91270; 307286
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Contraception; Hemostasis; Blood Coagulation
MeSH Terms: conditions — Thrombosis | interventions — drospirenone and ethinyl estradiol combination; drospirenone; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Yasmin (DRSP 3mg/EE 0.03 mg)
- Arm 2 (Active Comparator)
  Interventions: Drug: Microgynon (LNG 0.15 mg/EE 0.03 mg)

INTERVENTIONS:
Drug: Yasmin (DRSP 3mg/EE 0.03 mg) — The study medication was packaged in 21-tablet blister packs. Each subject kit contained 7 blister packs plus 1 reserve blister pack.Subjects randomly assigned to the treatment group received 21 consecutive days of hormonally active tablets (3mg DRSP/0.03 mgEE). In each treatment cycle 21 tablets (1 tablet daily) have to be taken in sequence, followed by a pill-free interval of 7 days. The treatment period was 7 cycles (28 days per cycle).
  Arms: Arm 1
Drug: Microgynon (LNG 0.15 mg/EE 0.03 mg) — The study medication was packaged in 21-tablet blister packs. Each subject kit contained 7 blister packs plus 1 reserve blister pack.Subjects randomly assigned to the treatment group received 21 consecutive days of hormonally active tablets (LNG 0.15 mg/EE 0.03 mg). In each treatment cycle 21 tablets (1 tablet daily) have to be taken in sequence, followed by a pill-free interval of 7 days. The treatment period was 7 cycles (28 days per cycle).
  Arms: Arm 2

SUMMARY:
The objective of this study was to investigate the impact of the oral contraceptive YASMIN (containing: drospirenone 3 mg/ethinyl estradiol 30 mcg) in comparison with the oral contraceptive MICROGYNON (containing: levonorgestrel 150 mcg/ethinyl estradiol 30mcg) on factors of blood coagulation and fibrinolysis in female subjects

ELIGIBILITY:
Inclusion Criteria:

* Clinically normal safety laboratory results

Exclusion Criteria:

* Standard contraindications for use of combined oral contraceptives (class label). Including:

  * Presence or history of thromboembolic process in veins (such as deep venous thrombosis, pulmonary embolism) or arteries (e.g., stroke, myocardial infarction) or a known genetic component (homozygous), venous thromboembolic event in a close relative (parents or siblings) at younger age (</= 40 years)
* Acute and chronic severe liver dysfunction or disease. There should be an interval of at least 6 months between the subsidence of a viral hepatitis (normalization of the liver parameters) and the start of the study medication.
* Use of preparations where experience shows affect on the activity of hepatic enzymes.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2003-06; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Pro-coagulatory parameters: Factor VIII (activity), Fibrinogen | At baseline and after wash out (period 2); after 7 cycles of treatment in each of the two study periods
Anti-coagulatory parameters: Protein C (activity), Antithrombin III(activity), APC resistance (factor V mutation) | At baseline and after wash out (period 2); after 7 cycles of treatment in each of the two study periods

SECONDARY OUTCOMES:
Rosing test: APC sensitivity ratio | At baseline and after wash out (period 2); after 7 cycles of treatment in each of the two study periods
Pro-coagulatory parameters: Factor VIII (activity), Activation markers: D-dimer, Prothrombin fragment 1+2 | At baseline and after wash out (period 2); after 7 cycles of treatment in each of the two study periods

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany